CLINICAL TRIAL: NCT00305864
Title: A PHASE I/II TRIAL OF TEMOZOLOMIDE, MOTEXAFIN GADOLINIUM, AND 60 GY FRACTIONATED RADIATION FOR NEWLY DIAGNOSED SUPRATENTORIAL GLIOBLASTOMA MULTIFORME
Brief Title: Motexafin Gadolinium, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01092; NCI-2009-01092 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000467802; RTOG 0513 (Other: Radiation Therapy Oncology Group); RTOG-0513 (Other: CTEP); U10CA021661 (NIH)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy, Conformal; motexafin gadolinium; Temozolomide

ARMS (4):
- Phase I: MGd 3 mg/kg (Experimental): Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning the night before the first dose of radiotherapy and ending the night before the last dose of radiotherapy, patients receive concurrent oral temozolomide once daily on days 0-39. Patients also receive MGd IV over 30 minutes prior to radiotherapy once daily on days 1-5 and 8-12 and then on days 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, and 40. Beginning 28 days after the completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Motexafin Gadolinium; Drug: Temozolomide
- Phase I: MGd 4 mg/kg (Experimental): Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning the night before the first dose of radiotherapy and ending the night before the last dose of radiotherapy, patients receive concurrent oral temozolomide once daily on days 0-39. Patients also receive MGd IV over 30 minutes prior to radiotherapy once daily on days 1-5 and 8-12 and then on days 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, and 40.Beginning 28 days after the completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Motexafin Gadolinium; Drug: Temozolomide
- Phase I: MGd 5 mg/kg (Experimental): Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning the night before the first dose of radiotherapy and ending the night before the last dose of radiotherapy, patients receive concurrent oral temozolomide once daily on days 0-39. Patients also receive MGd IV over 30 minutes prior to radiotherapy once daily on days 1-5 and 8-12 and then on days 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, and 40. Beginning 28 days after the completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5.Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Motexafin Gadolinium; Drug: Temozolomide
- Phase II: MGd 5 mg/kg (Active Comparator): Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning the night before the first dose of radiotherapy and ending the night before the last dose of radiotherapy, patients receive concurrent oral temozolomide once daily on days 0-39. Patients also receive MGd IV over 30 minutes prior to radiotherapy once daily on days 1-5 and 8-12 and then on days 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, and 40. Beginning 28 days after the completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Motexafin Gadolinium; Drug: Temozolomide

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo radiotherapy
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Drug: Motexafin Gadolinium — Given IV
  Other Names: API-GP3; gadolinium texaphyrin; Gd (III) Texaphryin; Gd-Tex; PCI-0120; Xcytrin
Drug: Temozolomide — Given orally
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase I/II trial is studying the side effects and best dose of motexafin gadolinium when given together with temozolomide and radiation therapy and to see how well they work in treating patients with newly diagnosed supratentorial glioblastoma multiforme or gliosarcoma. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Motexafin gadolinium may help temozolomide work better by making tumor cells more sensitive to the drug. Radiation therapy uses high-energy x-rays to kill tumor cells. Motexafin gadolinium may also make tumor cells more sensitive to radiation therapy. Giving motexafin gadolinium together with temozolomide and radition therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of motexafin gadolinium (MGd) when given concurrently with temozolomide and radiotherapy in patients with newly diagnosed supratentorial glioblastoma multiforme (GBM) or gliosarcoma.

II. Estimate the overall survival of patients treated with concurrent radiotherapy, temozolomide, and MGd followed by post-radiation temozolomide.

III. Determine the short- and long-term adverse effects in patients treated with this treatment.

IV. Estimate the progression-free survival of patients with newly diagnosed supratentorial GBM or gliosarcoma treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of motexafin gadolinium (MGd).

PHASE I: Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning the night before the first dose of radiotherapy and ending the night before the last dose of radiotherapy, patients receive concurrent oral temozolomide once daily on days 0-39. Patients also receive MGd IV over 30 minutes prior to radiotherapy once daily on days 1-5 and 8-12 and then on days 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, and 40. Beginning 28 days after the completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-7 patients receive escalating doses of MGd until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which no more than 6 eligible patients experience dose-limiting toxicity.

PHASE II: Patients undergo radiotherapy and receive temozolomide as in phase I. Patients also receive MGd as in phase I at the MTD determined in phase I.

After completion of study treatment, patients are followed every 2 months for 1 year, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme (GBM) or gliosarcoma

  * Newly diagnosed by surgical biopsy or excision within the past 5 weeks
* Supratentorial location, as determined by the following:

  * Contrast-enhanced MRI performed preoperatively
  * MRI performed postoperatively within 28 days prior to study entry (preferably within 72 hours of surgery)
  * Postoperative scan not required if diagnosed by stereotactic biopsy and pre-operative MRI was performed
* No gliomas graded < GBM
* No recurrent malignant gliomas
* No tumor foci detected below the tentorium or beyond the cranial vault
* No multifocal disease or leptomeningeal spread
* Zubrod performance status 0-1
* Neurologic function status 0-2
* Absolute neutrophil count ≥ 1,800 cells/mm^3
* Platelet count ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 8 g/dL (transfusion allowed)
* BUN ≤ 25 mg/dL
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* ALT or AST ≤ 2 times upper limit of normal
* Fertile patients must use effective contraception during and for 2 months after completion of study treatment
* Negative pregnancy test
* Not pregnant or nursing
* No prior invasive malignancies, except for nonmelanomatous skin cancer and carcinoma in situ of the uterine cervix or bladder, unless disease-free for ? 3 years
* No severe, active comorbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at study entry
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to study entry
  * Coagulation defects
  * Known AIDS
* No prior allergic reaction to the study drugs
* No history of porphyria or G6PD deficiency
* No allergy to gadolinium or contraindications to MRI
* No other concurrent chemotherapy
* Recovered from effects of surgery or postoperative infection and other complications
* No prior systemic chemotherapy, including polifeprosan 20 with carmustine implant (Gliadel wafer), for the current GBM

  * Prior chemotherapy for a different cancer allowed
* No prior radiotherapy to the head and neck (except for T1 glottic cancer) that would result in overlap of radiation therapy fields
* No prophylactic filgrastim (G-CSF) during the first course of study treatment
* No concurrent sargramostim (GM-CSF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-02-09 (Actual); Primary Completion 2011-02-16 (Actual); Study Completion 2011-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Brachman, Principal Investigator — Radiation Therapy Oncology Group
Locations (106):
- United States (106):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arizona Oncology Services Foundation, Scottsdale, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Saint Rose Hospital, Hayward, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Denver Veterans Administration Medical Center, Denver, Colorado
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Franciscan Saint Margaret Health-Hammond Campus, Hammond, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Mercy Hospital-Joplin, Joplin, Missouri
  - CHI Health Good Samaritan, Kearney, Nebraska
  - John F Kennedy Medical Center, Edison, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Washington Medical Center, Seattle, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Brachman DG, Pugh SL, Ashby LS, Thomas TA, Dunbar EM, Narayan S, Robins HI, Bovi JA, Rockhill JK, Won M, Curran WP. Phase 1/2 trials of Temozolomide, Motexafin Gadolinium, and 60-Gy fractionated radiation for newly diagnosed supratentorial glioblastoma multiforme: final results of RTOG 0513. Int J Radiat Oncol Biol Phys. 2015 Apr 1;91(5):961-7. doi: 10.1016/j.ijrobp.2014.12.050. PMID 25832688

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In multicenter clinical trials the accrual closure date must be predicted so that sites can be notified weeks in advance. As expected, this process often results in a final number of patients differing from the planned accrual.
Groups:
- Phase I: MGd 4 mg/kg; Phase I: MGd 5 mg/kg; Phase II: MGd 5 mg/kg: Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning the night before the first dose of radiotherapy and ending the night before the last dose of radiotherapy, patients receive concurrent oral temozolomide once daily on days 0-39. Patients also receive MGd IV over 30 minutes prior to radiotherapy once daily on days 1-5 and 8-12 and then on days 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, and 40. Beginning 28 days after the completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I: MGd 3 mg/kg | Phase I: MGd 4 mg/kg | Phase I: MGd 5 mg/kg | Phase II: MGd 5 mg/kg
Started | 7 | 10 | 7 | 94
Completed | 7 | 9 | 6 | 81
Not Completed | 0 | 1 | 1 | 13
Not completed — Ineligible / No protocol treatment | 0 | 1 | 1 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: MGd 3 mg/kg | Phase I: MGd 4 mg/kg | Phase I: MGd 5 mg/kg | Phase II: MGd 5 mg/kg | Total
Number analyzed (Participants) | 7 | 10 | 7 | 94 | 118
Age, Continuous [Median (Full Range); unit: years] | 56 [44 to 67] | 57.5 [37 to 72] | 58 [40 to 65] | 57.5 [20 to 81] | 57 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 1 | 33 | 44
  Male | 3 | 4 | 6 | 61 | 74

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of MGd (Phase I)
Description: Patients were to be followed for a minimum of 90 days from the start of radiation therapy (RT) and carefully evaluated with respect to treatment morbidity. A dose limiting toxicity (DLT) was defined as a grade 4 neurologic adverse event (AE) considered to be related to treatment occurring within 21 days of the conclusion of RT. For each dose level, up to seven patients were to be accrued to assure that there would be six eligible for treatment adverse event evaluation. A dose level of MGd was considered acceptable if no more than 1 patient of the 6 experience a DLT. If the current level was considered acceptable, then dose escalation occurred. Otherwise, the preceding dose level would be declared the maximum tolerated dose (MTD). The MTD would be used for the Phase II arm.
  Rating scale: 0 = not the MTD, 1 = MTD
Time Frame: From start of radiation therapy to 90 days,
Population: Eligible patients who received protocol treatment.
Measure: Number; unit: units on a scale
Groups:
- Phase I: 5 mg/kg: Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning the night before the first dose of radiotherapy and ending the night before the last dose of radiotherapy, patients receive concurrent oral temozolomide once daily on days 0-39. Patients also receive MGd IV over 30 minutes prior to radiotherapy once daily on days 1-5 and 8-12 and then on days 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, and 40. Beginning 28 days after the completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase I: MGd 3 mg/kg | Phase I: MGd 4 mg/kg | Phase I: 5 mg/kg
Number analyzed (Participants) | 7 | 9 | 6
units on a scale | 0 | 0 | 1

2. Primary Outcome: Median Overall Survival (Phase II)
Description: Survival time was defined as the time from baseline to date of death from any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for at least 18 months. Patients were followed up to 54.3 months
Population: All eligible patients.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- All MGd 5mg/kg Patients (Phase I and II Arms Combined): Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Beginning the night before the first dose of radiotherapy and ending the night before the last dose of radiotherapy, patients receive concurrent oral temozolomide once daily on days 0-39. Patients also receive MGd IV over 30 minutes prior to radiotherapy once daily on days 1-5 and 8-12 and then on days 15, 17, 19, 22, 24, 26, 29, 31, 33, 36, 38, and 40. Beginning 28 days after the completion of radiotherapy, patients receive oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | All MGd 5mg/kg Patients (Phase I and II Arms Combined)
Number analyzed (Participants) | 87
Months | 15.6 [12.9 to 17.6]
Statistical Analysis 1: Comparison: All MGd 5mg/kg Patients (Phase I and II Arms Combined); A one-sided one-sample log-rank test at significance level of 0.10 was predicted to have 85% power to detect a survival difference against the historical control (13.7 vs. 18.5 months) with 60 deaths; Test type: Superiority or Other; p = 0.27, Log Rank; One-sided

3. Secondary Outcome: Progression-free Survival (Phase II)
Description: Progression will be defined as a > 25% increase in tumor area. Progression-free survival time was defined as the time from baseline to date of death from any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: From randomization to date of progression, death, or last follow-up. Analysis occurs after all patients have been potentially followed for at least 18 months. Patients were followed up to 54.3 months.
Population: All eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All MGd 5mg/kg Patients (Phase I and II Arms Combined)
Number analyzed (Participants) | 87
months | 7.6 [5.7 to 9.6]

ADVERSE EVENTS:
Description: Per the protocol, toxicity data was collected via Common Toxicity Criteria (CTC) 3.0 then mapped to CTCAE 4.0 for reporting on this website. Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. Subjects experiencing more than one of a given "Other (Not Including Serious)" adverse event (AE) are counted only once for that "Other (Not Including Serious)" AE.
Arm/Group | Phase I: MGd 3 mg/kg | Phase I: MGd 4 mg/kg | Phase I: MGd 5 mg/kg | Phase II: MGd 5 mg/kg
Serious Adverse Events (participants affected / at risk) | 3/7 | 6/9 | 4/6 | 48/81
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9 | 6/6 | 80/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: MGd 3 mg/kg (N=7) | Phase I: MGd 4 mg/kg (N=9) | Phase I: MGd 5 mg/kg (N=6) | Phase II: MGd 5 mg/kg (N=81)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 3
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 4
Death NOS (General disorders) | 0 | 0 | 0 | 2
Edema limbs (General disorders) | 0 | 0 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 11
Fever (General disorders) | 0 | 0 | 1 | 12
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Sudden death NOS (General disorders) | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 4
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 1 | 4
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1
Phlebitis infective (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 7
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 5
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 9
Neutrophil count decreased (Investigations) | 1 | 3 | 0 | 6
Platelet count decreased (Investigations) | 1 | 2 | 0 | 7
White blood cell decreased (Investigations) | 1 | 2 | 0 | 10
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 2 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 2
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 2
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 4
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 2
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 4
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Thromboembolic event (Vascular disorders) | 0 | 2 | 1 | 4
Vascular disorders - Other (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: MGd 3 mg/kg (N=7) | Phase I: MGd 4 mg/kg (N=9) | Phase I: MGd 5 mg/kg (N=6) | Phase II: MGd 5 mg/kg (N=81)
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 2 | 41
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 0 | 3
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 3
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 3
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 2 | 5
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 6
Cushingoid (Endocrine disorders) | 0 | 1 | 0 | 2
Endocrine disorders - Other (Endocrine disorders) | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 1 | 1 | 2 | 13
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 4
Extraocular muscle paresis (Eye disorders) | 0 | 0 | 1 | 4
Eye disorders - Other (Eye disorders) | 4 | 0 | 1 | 20
Eye pain (Eye disorders) | 0 | 1 | 0 | 2
Flashing lights (Eye disorders) | 0 | 0 | 1 | 1
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 1 | 0 | 2
Uveitis (Eye disorders) | 0 | 0 | 1 | 0
Watering eyes (Eye disorders) | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Anal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 3 | 2 | 39
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 1 | 20
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastric stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Nausea (Gastrointestinal disorders) | 4 | 2 | 3 | 55
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0 | 28
Chills (General disorders) | 0 | 1 | 0 | 15
Death NOS (General disorders) | 0 | 0 | 0 | 1
Edema face (General disorders) | 0 | 0 | 0 | 3
Edema limbs (General disorders) | 3 | 1 | 0 | 16
Edema trunk (General disorders) | 1 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 6 | 7 | 5 | 70
Fever (General disorders) | 0 | 1 | 0 | 15
Flu like symptoms (General disorders) | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 5
General disorders and administration site conditions - Other (General disorders) | 1 | 0 | 0 | 4
Injection site reaction (General disorders) | 0 | 3 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 2 | 8
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0 | 3 | 11
Bladder infection (Infections and infestations) | 0 | 1 | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1
Gum infection (Infections and infestations) | 0 | 0 | 1 | 3
Infections and infestations - Other (Infections and infestations) | 1 | 1 | 0 | 9
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 3
Vulval infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 6
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 3 | 2 | 16
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 4 | 4 | 49
Alkaline phosphatase increased (Investigations) | 1 | 3 | 0 | 19
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 2 | 34
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 8
Cholesterol high (Investigations) | 0 | 0 | 0 | 1
Creatinine increased (Investigations) | 1 | 1 | 0 | 10
GGT increased (Investigations) | 0 | 0 | 0 | 4
Haptoglobin decreased (Investigations) | 0 | 1 | 0 | 0
INR increased (Investigations) | 1 | 1 | 0 | 0
Investigations - Other (Investigations) | 3 | 1 | 1 | 11
Lipase increased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 3 | 1 | 47
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 14
Platelet count decreased (Investigations) | 2 | 3 | 2 | 37
Serum amylase increased (Investigations) | 0 | 0 | 0 | 1
Weight gain (Investigations) | 0 | 1 | 0 | 4
Weight loss (Investigations) | 2 | 1 | 1 | 19
White blood cell decreased (Investigations) | 1 | 1 | 0 | 32
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 3 | 4 | 37
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 3 | 0 | 36
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 19
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 29
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 5
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 7 | 3 | 56
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 24
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 10
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 12
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 7
Acoustic nerve disorder NOS (Nervous system disorders) | 0 | 0 | 1 | 3
Ataxia (Nervous system disorders) | 0 | 1 | 1 | 5
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 0 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 5
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 6
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 12
Dysgeusia (Nervous system disorders) | 4 | 2 | 3 | 19
Dysphasia (Nervous system disorders) | 1 | 2 | 2 | 8
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 2
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 2 | 2 | 45
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 2
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 1 | 21
Nervous system disorders - Other (Nervous system disorders) | 0 | 0 | 0 | 6
Neuralgia (Nervous system disorders) | 2 | 2 | 1 | 5
Oculomotor nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 1 | 18
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2 | 2 | 27
Seizure (Nervous system disorders) | 1 | 3 | 2 | 11
Sinus pain (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 8
Agitation (Psychiatric disorders) | 0 | 1 | 2 | 6
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 15
Confusion (Psychiatric disorders) | 0 | 1 | 3 | 22
Depression (Psychiatric disorders) | 1 | 1 | 1 | 14
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 21
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 1 | 15
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urine discoloration (Renal and urinary disorders) | 5 | 3 | 2 | 25
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5 | 4 | 56
Body odor (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 10
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Nail loss (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 15
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 17
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 14
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 13
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 31
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 | 5 | 2 | 33
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Flushing (Vascular disorders) | 0 | 1 | 2 | 4
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1 | 13
Hypotension (Vascular disorders) | 0 | 1 | 1 | 3
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 3 | 0 | 3
Vascular disorders - Other (Vascular disorders) | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less